CLINICAL TRIAL: NCT02992470
Title: Hydrolyzed Oyster Extract for Liver Health: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Crassostrea Gigas for Liver Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016_11_Crassostrea gigas
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrolyzed oyster extract (Experimental): A 250 mg, film-coated oblong (rectangle) shaped tablet of oyster extract
  Interventions: Dietary Supplement: Hydrolyzed oyster extract
- Placebo (Placebo Comparator): A 250 mg, film-coated oblong (rectangle) shaped tablet of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed oyster extract — 1 tablet of oyster extract t.i.d. for 8 weeks
  Arms: Hydrolyzed oyster extract
Dietary Supplement: Placebo — 1 tablet of maltodextrin t.i.d. for 8 weeks
  Arms: Placebo

SUMMARY:
This study aimed to observe whether a hydrolyzed oyster extract improves liver health in participants whose alanine transaminase (ALT) levels are1-3 fold above the normal. A total of 96 participants will be randomly allocated to active (oyster) or placebo group (1:1). Each group will receive 750 mg of oyster extract or placebo per day for 8 weeks. Primary outcome will be the change in ALT level and secondary outcomes will be; (1) ratios of participants with normal ALT, aspartate aminotransferase (AST), and gamma-glutamyl transferase (GGT); (2) the change in serum bilirubin; (3) the change in multi-dimensional fatigue inventory; (4) the changes in serum lipids; (5) the changes in antioxidant enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19
* AST, ALT, and GGT levels above the upper limit of the normal but less than 3 times the upper limit of the normal
* Participants with normal physical activity who sign an informed consent form
* Fatty liver detected by ultrasound

Exclusion Criteria:

* Allergic reaction to oyster
* Uncontrolled diabetes mellitus
* Active viral hepatitis and any liver diseases that can affect trial outcomes (positive for HBs Ag or HCV Ab)
* Liver cirrhosis of Child-Pugh class B or C
* Chemotherapy or radiation therapy for cancer within 6 months
* Cholelithiasis
* Systemic medications that can affect liver function such as INH, valproic acid, tetracycline, allopurinol, phenytoin, phenelzine, sertraline, naproxen and diclofenac within 4 weeks
* Medication of cholagogues, cholelitholytics & hepatic protectors, antidotes, detoxifying agents, and drug abuse (drugs used in substance dependence) within 4 weeks
* Alcoholism or excessive alcohol intake of more than 168 g/week in men and 112 g/week in women
* Kidney diseases or serum creatinine level above 2.0 mg/dL
* Uncontrolled hypertension or angina pectoris or myocardiac infarction
* History of bowel resection (not including surgery on simple appendicitis)
* Medication of antipsychotic drugs
* Herbal medication within 2 months
* Pregnancy or breastfeeding
* Participation of other clinical trial(s) within 1 months from screening day
* Uncooperativeness
* Intake of dietary supplements within 4 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of serum alanine aminotransferase (ALT) | Baseline, 4 weeks and 8 weeks

SECONDARY OUTCOMES:
Change of serum aspartate aminotransferase (AST) | Baseline, 4 weeks and 8 weeks
Change of gamma-glutamyl transferase (GGT) | Baseline, 4 weeks and 8 weeks
Rate of participants with normalized ALT, AST and GGT | Baseline, 4 weeks and 8 weeks
Change of serum bilirubin | Baseline, 4 weeks and 8 weeks
Change of multi-dimensional fatigue inventory | Baseline, 4 weeks and 8 weeks
Change of serum lipid profiles (triglyceride, total cholesterol, High-density lipoprotein and low-density lipoprotein cholesterol) | Baseline, 4 weeks and 8 weeks
Change of antioxidant enzymes (superoxide dismutase, malondialdehyde, glutathione peroxidase) | Baseline, 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Yong Choi, Principal Investigator — Korean Medicine Hospital, Pusan National University